CLINICAL TRIAL: NCT07113184
Title: DUAL VERSUS SINGLE STENTRIEVER FOR RECANALIZATION IN ACUTE ISCHEMIC STROKE: THE RANDOMIZED DOUBLE UP TRIAL
Brief Title: Randomized a Clinical Trial With Medical Device in Acute Ischemic Stroke
Acronym: DOBLE UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOBLE UP
Record Dates: First submitted 2025-07-11; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; mechanical thrombectomy; dual stentriever; mTICI; first pass effect; randomized trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Endovascular mechanical thrombectomy with either dual or single stentriever technique using a balloon guiding catheter.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Stentriever (Experimental): Endovascular mechanical thrombectomy with dual or stentriever technique using a balloon guiding catheter.
  Interventions: Device: dual sr
- Single Stentriever (Active Comparator): Endovascular mechanical thrombectomy with single stentriever technique using a balloon guiding catheter.
  Interventions: Device: single sr

INTERVENTIONS:
Device: dual sr — Dual Stentriever
  Other Names: experimental
  Arms: Dual Stentriever
Device: single sr — Single Stentriever
  Other Names: control
  Arms: Single Stentriever

SUMMARY:
This study seeks to provide high-quality evidence on the potential benefits of the dual stentriever approach, potentially informing future clinical guidelines and improving outcomes in patients with anterior circulation large vessel occlusion strokes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* NIHSS ≥ 6
* mRS ≤ 1
* Proximal anterior circulation occlusion
* ASPECTS > 6
* Informed consent

Exclusion Criteria:

* Absence of occlusion
* Posterior circulation stroke
* Carotid dissection or tandem stenosis requiring treatment
* Severe comorbidities or contraindications to imaging contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time takes in achieving complete reperfusion after a single thrombectomy pass. | 24 hours or 48 hours after thrombectomy
  To evaluate the superiority of the dual stentriever technique in achieving complete reperfusion after a single thrombectomy pass.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital de Burgos, Burgos
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital universitario marques de valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No